CLINICAL TRIAL: NCT01056133
Title: A Pilot Study to Determine the Effect of Omega-3 Polyunsaturated Fatty Acids From Fish Oil on Patients With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Effect of Fish-oil on Non-alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johane Allard (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); American College of Gastroenterology (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Professor, Gastroenterologist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0874-A; CIHR Grant#89705 (Other Grant/Funding Number: Canadian Institutes of Health Research); MOP-123459 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: non-alcoholic fatty liver disease; non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 capsules-Fish Oil (Experimental): Omega-3 fatty acids in the form of fish oil capsules (2g/d)
  Interventions: Other: Omega-3 capsules-Fish Oil

INTERVENTIONS:
Other: Omega-3 capsules-Fish Oil — Patients will take 2 capsules (1.0 g each) of n-3 PUFA (0.82/0.44 g of EPA/DHA) daily x 12 months. Since n-3 PUFA supplementation can be a potential treatment for NASH and since BMI will be< 30 kg/m2 for all subjects, patients will be told to keep their lifestyle, diet and medication stable (unless medically necessary) for the study duration in order to minimize environmental effect on gene expression.
  Other Names: Product Name: Amber 40/20 Ethyl ester (EE); 1000 mg capsules (lemon-lime flavor); Product Code: 4020PB1000CT

SUMMARY:
The purpose of this study is to determine the effect of Omega-3 Fish oil supplementation on hepatic gene expression in patients with Non Alcoholic Steatohepatitis (NASH). In addition, effects of fish oil on intestinal microbiota will be assessed.

DETAILED DESCRIPTION:
Changes in fatty acid (FA) composition within the liver may influence lipid metabolism and inflammation. This is poorly understood in humans.

Especially omega-3 FA are important: They promote FA oxidation over storage and are important for export of lipids from the liver. Omega-3 FA have also anti-inflammatory properties.

Changes in liver FA composition may be influenced by dietary intake, high rate of lipid peroxidation (LP) or low delta-6 desaturase enzyme activity. We and others recently showed that NASH patients had lower hepatic n-3 and n-6 polyunsaturated FA (PUFA) with increased lipid peroxidation and low antioxidant status when compared to patients with minimal findings on liver biopsy. The dietary intake of FA was similar among the 3 groups suggesting that the difference in hepatic FA composition may be related to high lipid peroxidation or low delta-6 desaturase activity. This difference in hepatic FA composition may be of significance in the pathogenesis of NASH since it may change gene expressions in regard to lipid metabolism.

This pilot study in NASH to assess the effect of n-3 PUFA supplementation on FA composition (liver and red blood cells), hepatic gene expression, and histology. We will also assess the ratio of phosphatidylcholine (PC) to phosphatidylethanolamine (PE) in liver and red blood cells (RBC). Oxidative stress, insulin resistance and nutritional measurements will be performed to further characterize these patients.

New research suggests that the composition of the gut flora (intestinal microbiota) may play a role in the development of NASH. The effect of fish oil on the intestinal microbiota has not been examined in humans. Therefore, intestinal microbiota is also measured before and after intervention and associations between changes in microbiota and changes in liver histology will be examined. In addition, bacterial products (short chain fatty acids in stool, lipopolysaccharide in plasma, bacterial DNA in plasma), and plasma choline will be measured. An environmental questionnaire will capture factors that can influence the intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven NASH; male and female; age 18-65 years; BMI ≤ 40 kg/m2, alcohol consumption <20g/d; non-smokers; if known to have hyperlipidemia or diabetes, need to be stable drug regimen.

Exclusion Criteria:

* Liver disease of other etiology; documented HIV infection, anticipated need for liver transplantation in one year or complications such as recurrent variceal bleeding, spontaneous portosystemic encephalopathy, ascites or jaundice; concurrent medical illnesses, abnormal coagulation or other reasons judged by the hepatologist to contraindicate a liver biopsy; chronic gastrointestinal diseases, previous gastrointestinal surgery modifying the anatomy, patients with diabetes requiring insulin; medications known to precipitate steatohepatitis in the 6 months prior to entry; regular intake of non-steroidal anti-inflammatory drugs, regular intake of antioxidant vitamin or omega-3/fish oil supplements, prebiotics, probiotics, antibiotics, or laxatives; ursodeoxycholic acid or any experimental drug in the 6 months prior to study entry; smokers; pregnancy or lactating; female subjects who are not surgically sterile or postmenopausal and who are not using medically acceptable methods of birth control during the trial and for 30 days after the treatment period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Liver histology | Baseline, 12 months
  Liver histology will be assessed for diagnosis of NASH (steatosis, inflammation, ballooning, fibrosis, mallory bodies, Non-alcoholic fatty liver disease activity score (NAS)

SECONDARY OUTCOMES:
Plasma and RBC fatty acid composition and PC:PE ratio | At 3,6,12 months
Blood biochemistry (blood sugar control, lipid profile, liver enzymes) | Baseline, 6, 12 months
Intestinal microbiota | Baseline, 6, 12 months
  Composition of intestinal microbiota will be measured in stool samples using Ion Torrent technology and quantitative reverse transcription polymerase chain reaction
Plasma endotoxin | Baseline, 6, 12 months
Plasma free choline | Baseline, 6, 12 months
Bacterial DNA in plasma | Baseline, 6, 12 months

OTHER OUTCOMES:
Environmental questionnaire | Baseline, 6, 12 months
  To assess factors that influence intestinal microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada